CLINICAL TRIAL: NCT03645772
Title: Plyometric Exercise to Improve Rapid Force Production in Older Men: a Pilot Intervention
Brief Title: Plyometric Exercise to Improve Rapid Force Production in Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Evelien Van Roie, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S60983
Record Dates: First submitted 2018-08-17; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Exercise Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plyometric exercise (Experimental): 12-week progressive exercise program, consisting of plyometric exercises such as countermovement jump, forward and sideways step-up.
  Interventions: Other: Exercise intervention
- Resistance exercise (Active Comparator): 12-week resistance exercise program for the leg muscles (2-4 sets of 8-15 repetitions at 8-15RM, leg press, leg extension, calve extension).
  Interventions: Other: Exercise intervention
- Walking (Active Comparator): 12-week progressive walking program.
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — 12-week progressive training intervention

SUMMARY:
Rapid force production declines as a consequence of ageing. Given the functional relevance of rapid force production, exercise interventions in older adults should aim at improving the capacity to produce force rapidly. To improve this capacity, exercises should be performed with the intention to develop high speeds, as supported by previous work.

Human locomotion fundamentally consists of multi-joint movements and rapidly coupled eccentric-concentric muscle actions, known as stretch-shortening cycle (SSC) activities or plyometrics. Plyometrics might therefore be used to optimize power production. However, there is limited research on the feasibility of plyometrics in older adults and its potential effects on rapid force production and functional capacity. This study will test the feasibility of a 12-week plyometric exercise intervention in older men and compare its effects on rapid force production to a traditional resistance exercise or walking intervention.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* No systematic engagement in (resistance) exercise in the 12-months prior to participation
* Cardiovascular disease
* Neurological disorders
* Cognitive malfunctioning
* Severe knee or hip problems

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Rapid force production | Change from baseline in rapid force production at 12 weeks
  Subjects perform a test protocol on a sledge apparatus, consisting of explosive isometric voluntary contractions for the leg-extensor muscles of the right leg. The inclination of the sledge is 20° to horizontal. The seat of the sledge is inclined backwards (130°). The knee joint angle is set at 90° and the hip angle at 70°. The point of force application is aligned with the head of the fifth metatarsal. Subjects are instructed to kick as fast and as hard as possible and maintain their maximum force for approximately 3s. The rate of force development (N/s) is defined as the linear slope of the force-time curve and is measured from the onset of movement till 100 ms.
Jumping height in squat jump | Change from baseline in jumping height at 12 weeks
  Subjects perform a test protocol on a sledge apparatus, consisting of squat jumps (SJ), countermovement jumps (CMJ), and drop jumps (DJ). The inclination of the sledge is 20° to horizontal. The seat of the sledge is inclined backwards (130°). A force platform is built in perpendicular to the jumping direction. A speed sensor is attached to the seat of the sledge, which is used to assess the transition point between braking and push-off phases and to calculate jumping height (in cm).
Jumping height in countermovement jump | Change from baseline in jumping height at 12 weeks
  Subjects perform a test protocol on a sledge apparatus, consisting of squat jumps (SJ), countermovement jumps (CMJ), and drop jumps (DJ). The inclination of the sledge is 20° to horizontal. The seat of the sledge is inclined backwards (130°). A force platform is built in perpendicular to the jumping direction. A speed sensor is attached to the seat of the sledge, which is used to assess the transition point between braking and push-off phases and to calculate jumping height (in cm).
Jumping height in drop jump | Change from baseline in jumping height at 12 weeks
  Subjects perform a test protocol on a sledge apparatus, consisting of squat jumps (SJ), countermovement jumps (CMJ), and drop jumps (DJ). The inclination of the sledge is 20° to horizontal. The seat of the sledge is inclined backwards (130°). A force platform is built in perpendicular to the jumping direction. A speed sensor is attached to the seat of the sledge, which is used to assess the transition point between braking and push-off phases and to calculate jumping height (in cm).

SECONDARY OUTCOMES:
Leg press one-repetition maximum | Change from baseline in leg press 1-RM at 12 weeks
  Leg press one-repetition maximum is defined as the maximum weight (in kg) that the subject can push on a leg press device (Signature Series Leg press Life Fitness).
Maximal isometric strength | Change from baseline in maximal isometric strength at 12 weeks
  Maximal strength (Nm) is measured by means of unilateral isometric knee-extensor tests on a Biodex dynamometer.
Maximal isokinetic strength | Change from baseline in maximal isokinetic strength at 12 weeks
  Maximal strength (Nm) is measured by means of unilateral isokinetic knee-extensor tests on a Biodex dynamometer.
Stair Climbing performance | Change from baseline in Stair Climbing performance at 12 weeks
  Stair ascent duration (in s), the time needed to ascent a flight of stairs.
Gait speed | Change from baseline in gait speed at 12 weeks
  The average speed to walk 10m as fast as possible (in m/s).
5 repetition sit-to-stand test | Change from baseline in sit-to-stand duration at 12 weeks
  The time needed to perform 5 sit-to-stand transitions (in s).
6 minute walk distance | Change from baseline in 6min walk distance at 12 weeks
  The walk distance (in m) covered in 6 min.
Balance | Change from baseline in balance at 12 weeks
  Overall balance performance is assessed using the total length of the sway path divided by duration of the measurement (mm/s) in a 30s balance test on a balance board.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Movement Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No